CLINICAL TRIAL: NCT03838640
Title: Feasibility of Transnasal ECHO for Identification of Parapharyngeal Internal Carotid Artery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Arkadi Yakirevitch, Principal Investigator, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 5450-18-SMC
Record Dates: First submitted 2018-12-24; First posted 2019-02-12 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: To Assess Feasibility of the New Application

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study group (Experimental): Consecutive eligible patients requiring endoscopic surgery for sinonasal pathology Transnasal localization of internal carotid artery with TEE ECHO device will be performed
  Interventions: Device: EPIQ 5

INTERVENTIONS:
Device: EPIQ 5 — As described in summary Trade name of the device Philips EPIQ 5

SUMMARY:
Identification and preservation of internal carotid artery during endoscopic nasopharyngectomy in cases of malignancy is a main difficulty of this kind of surgery, especially when anatomy is distorted by previous radiation. Intraoperative navigation based on preoperative imaging cannot remain precise throughout the process of resection. We aim to check a feasibility of internal carotid artery localization with the help of transnasal ultrasonic scanning. The most appropriate for this method existing device is an echocardiography system with pediatric transesophageal transducer.

We plan to use it in 20 patients undergoing elective surgery for inflammatory sino-nasal disease. After initiatioin of general anesthesia and local decongestion, transducer will be placed transnasally to nasopharynx in order to scan a parapharyngeal space.

ELIGIBILITY:
Inclusion Criteria:

Indication for endoscopic nose and paranasal sinuses surgery

Exclusion Criteria:

Previous nasopharyngeal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
distance from nasopharynx surface to a closest wall of internal carotid arter | 3 minutes
  cm

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No
No plans to share